

FOR IRB USE ONLY IRB ID #: 201912100 APPROVAL DATE: 01/20/22 RELEASED DATE: 01/20/22 EXPIRATION DATE: 01/19/23

De-Implementation of Unnecessary Surgical Antibiotic Prophylaxis in Children

We invite you to participate in a research study being conducted by [INSERT PI NAME] from [INSERT SITE NAME]. You are being asked to participate because you are an ASP or surgical team member.

In this proposed study, our multidisciplinary team will develop and test two theoretically informed strategies to eliminate ("de-implement") unnecessary postoperative antibiotic prophylaxis through the collaboration of surgeons and antimicrobial stewardship programs (ASPs) at approximately 10 centers across the United States. One promising strategy is the implementation of standard surgical order sets, which offer relative ease of implementation and a systematic approach across surgical subspecialties. While evidence suggests that order set standardization is a good approach, barriers to implementation are commonly noted. The purpose of this study is to develop, complementary strategies to extend the impact of order set standardization. The Agency for Healthcare Research and Quality is providing funding for this research study

If you agree to participate, you would need to complete several surveys either on-line or on paper at various time points over the next several years. If you do not want to participate in this study, please return the blank survey to us or exit the online survey. We will keep the information you provide confidential by removing any identifying information and using an ID code number instead of your name.

There are no known risks from being in this study, and you will not benefit personally. However, we hope that others may benefit in the future from what we learn as a result of this study.

You will not have any costs for being in this research study nor will you be paid for being in this research study.

We will keep the information you provide confidential by assigning a unique site and participant ID code number. The master list linking the ID codes to the sites/participants will be kept by the coordinating center and will be destroyed at the completion of all study activities. However, federal regulatory agencies and Washington University, including the Washington University Institutional Review Board (a committee that reviews and approves research studies) and the Human Research Protection Office may inspect and copy records pertaining to this research. If we write a report about this study we will do so in such a way that you cannot be identified.

• Identifiers may be removed from your private information and used for future research or shared with others. If this occurs, we will not ask you for additional consent.



FOR IRB USE ONLY IRB ID #: 201912100 APPROVAL DATE: 01/20/22 RELEASED DATE: 01/20/22 EXPIRATION DATE: 01/19/23

You will not have any costs for being in this research study.

You will not be paid for being in this research study.

Your participation in this study is completely voluntary. You may choose not to take part at all. If you decide to participate in the study you may stop participating at any time. Any data that was collected as part of this study will remain as part of the study records and cannot be removed. If you decide not to take part in the study or if you stop participating at any time, you won't be penalized or lose any benefits for which you otherwise qualify. We encourage you to ask questions. If you have questions for the research team, please contact [site name(s), phone number(s)]. If you feel you have been harmed from being in the study, please contact: [site name(s), phone number(s)] If you have questions, concerns, or complaints about your rights as a research participant, please contact the Human Research Protection Office at 1-(800)-438-0445 or email hrpo@wustl.edu. General information about being a research participant can be found on the Human Research Protection Office web site, <a href="http://hrpo.wustl.edu">http://hrpo.wustl.edu</a>. To offer input about your experiences as a research participant or to speak to someone other than the research staff, call the Human Research Protection Office at the number above.

Thank you very much for your consideration of this research study.

[Insert name of PI or Research Team Member] [Insert Title]